CLINICAL TRIAL: NCT01130636
Title: An Observational Study on the Pharmacokinetics of Oseltamivir in the Treatment of Influenza During Lactation, Phase IV Trial
Brief Title: Observational Study on the Pharmacokinetics of Oseltamivir in the Treatment of Influenza During Lactation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmahungary Group (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MV22970
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Influenza
Keywords: oseltamivir carboxylate; oseltamivir phosphate; Tamiflu pharmacokinetics in lactating women with influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir; Hardness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamiflu (Experimental): Lactating women (up to 20 subjects) who present with clinical symptoms indicative of influenza will be recruited (a maximum of 6 months period of recruitment) to receive immediate treatment with oseltamivir (Tamiflu® 75 mg hard capsules, provided free of charges for the study) at a standard dose of 75 mg twice daily. These subjects will have a 12 hour pharmacokinetic plasma, urine and breast milk study undertaken after the steady state in oseltamivir concentrations (both active and inactive metabolites will be measured) is reached in blood, i.e. after three days after treatment.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Lactating women who present with clinical symptoms indicative of influenza will receive immediate treatment with oseltamivir (Tamiflu® 75 mg hard capsules) at a standard dose of 75 mg twice daily.
  Other Names: Tamiflu® 75 mg hard capsules

SUMMARY:
The main purpose of this study is to assess the potential exposure of neonates to oseltamivir during lactation by examining oseltamivir concentrations in maternal blood, urine, and breast milk in breastfeeding women who are treated with oseltamivir, an anti-flu medication.

DETAILED DESCRIPTION:
Investigational Medical Product: Tamiflu® 75 mg hard capsules

Objective: The main purpose of this study is to assess the potential neonatal exposure to oseltamivir during lactation by examining oseltamivir concentrations in maternal blood, urine, and breast milk/colostrum.

Study design: Single-country, multicenter, observational pharmacokinetic study

Enrolment and follow-up: Lactating women (up to 20 subjects) who present with clinical symptoms indicative of influenza will be recruited (a maximum of 6 months period of recruitment) to receive immediate treatment with oseltamivir (Tamiflu® 75 mg hard capsules, provided free of charges for the study) at a standard dose of 75 mg twice daily. These subjects will have a 12 hour pharmacokinetic plasma, urine and breast milk study undertaken after the steady state in oseltamivir concentrations (both active and inactive metabolites will be measured) is reached in blood, i.e. after three days after treatment. Subjects do not need laboratory confirmation of influenza infection for inclusion in this study, although the results of any virological tests that seek to confirm influenza infection will be recorded. Maternal venous blood (2 samples, one pre-dose sample and one 2.5-hours-after-dose sample), urine samples (obtained from total urine output within 12 h), and breast milk/colostrum samples (8 samples within 12 h) are taken to determine oseltamivir phosphate (inactive metabolite) and oseltamivir carboxylate (active metabolite) levels.

Safety: Adverse events (AEs) and serious adverse events (SAEs) will be recorded. SAEs will be reported to the Ethics Committee and Regulatory authorities according to the reporting requirements in Hungary.

Number of patients: A total of 20 lactating patients will be enrolled.

Number of centres: Up to 3 investigational sites in Hungary will participate in the study. All sites will belong to an academic institution.

According to the approved protocol amendment 1 (dated: 31/Aug/2010) the time schedule is the following: The patient visits are planned as soon as possible during the pandemic season in Q3-Q4 2010 and Q1-Q2 2011. The study will run until enrollment is completed and all study procedures have been completed for the last subject in 2011.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is breastfeeding, or has just given birth.
2. The age of the patient is at least 18 years.
3. Written Informed Consent obtained from the patient.
4. The patient has received a diagnosis of influenza based upon the following clinical symptoms, during a time when influenza is known to be circulating:

   * fever ≥37.8oC at the time of examination or a history of fever and
   * at least one respiratory symptom (cough, coryza, sore throat, rhinitis)
5. Confirmation of infection with influenza is not required for inclusion. As H1N1v infection in pregnancy and lactation is a dangerous condition, and recommendations are that clinicians should commence antiviral therapy on an empiric basis and not wait for the results for laboratory investigations. Therefore, this study will not undertake or require any virological investigations, although these will be recorded if undertaken as part of routine care.

Exclusion Criteria:

1. Clinical suspicion of infection with a respiratory virus other than influenza and a decision by the treating physician that treatment with oseltamivir is not indicated.
2. Suspicion of invasive bacterial infection requiring immediate admission to hospital.
3. Evidence of a poorly controlled underlying medical condition, with the specific understanding that pregnancy does constitute an exclusion factor in this influenza-related study. Positive test with one of the following methods for pregnancy excludes patient from participation:

   * β-HCG blood test
   * β-HCG urine test
   * ultrasound examination confirming pregnancy.
4. Known or suspected immunosuppression (malignancy, transplant, immunosuppressive drugs)
5. Known allergy to oseltamivir.
6. Participation in any clinical trials with an investigational drug or vaccine within the previous 3 months.
7. A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the Investigator to be clinically significant and adversely affecting compliance to study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Oseltamivir phosphate and oseltamivir carboxylate concentration in venous blood, breast milk/colostrums, and urine. | 12 hour period
  For lactating women, the plasma concentrations of oseltamivir phosphate and oseltamivir carboxylate in venous blood, breast milk/colostrums, and urine measured over a 12 hour period after three days after treatment, when the steady state in oseltamivir concentrations (both active and inactive metabolites) is reached in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Vadász, MD, Principal Investigator — Selye János Hospital, Department of Obstetric and Gynecology,Komárom, Széchényi u.2. H-2921, Hungary; Tamás Major, MD PhD, Principal Investigator — DEOEC University of Debrecen, Clinic of Obstetrics and Gynecology, Debrecen, Nagyerdei krt. 98. H-4032, Hungary; Attila Pál, MD PhD DSc, Principal Investigator — Szeged University, Faculty of Medicine Szent-Györgyi Albert Clinical Center Clinic of Obstetrics and Gynecology; Nándor Ács, MD PhD, Principal Investigator — Semmelweis University II. Clinic of Obstetrics and Gynecology
Locations (2):
- Hungary (2):
  - DEOEC University of Debrecen, Clinic of Obstetrics and Gynecology, Debrecen
  - Selye János Hospital, Department of Obstetrics and Gynecology, Komárom